CLINICAL TRIAL: NCT07129486
Title: Intermittent-Hypoxia Inhibits Neutrophil Extracellular Traps Formation: Role of Cathelicidins
Status: Not yet recruiting | Type: Observational
Sponsor: Kun-Ta Chou (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Kun-Ta Chou, Chief, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Other Study IDs: 2025-02-007BC
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: sleep apnea; intermittent hypoxia; neutrophil extracellular traps; cathelicidins
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/Plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA: participants with OSA
  Interventions: Device: CPAP
- Control: Participants without OSA

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure (CPAP) is the standard treatment for moderate to severe OSA in clinical practice.
  Groups: OSA

SUMMARY:
The study will enroll 80 moderate-to-severe Obstructive sleep apnea (OSA) patients (40 obese) and 40 age-, gender-, and body mass index-matched controls. Venous blood will be collected to isolate neutrophils, which will be tested for the ability to produce neutrophil extracellular traps (NETs) along with the levels of LL-37 and NETs products in the blood. Measurements will be repeat after three months treatment for OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive upper airway collapse during sleep, thereby leading to intermittent hypoxia (IH). Literature revealed OSA confers a higher risk for poor infection outcomes, suggestive of defective immunity in those patients. This research aimed to investigate whether IH inhibits neutrophils to produce neutrophil extracellular traps (NETs) via Cathelicidins (LL-37). The human study will enroll 80 moderate-to-severe OSA patients (40 obese) and 40 age-, gender-, and body mass index-matched controls. Venous blood will be collected to isolate neutrophils, which receive either IH treatment (1% O2 for 35 mins and 21% for 25 mins per cycle, 3 cycles) or normoxic treatment. The neutrophils will be tested for the ability to produce NETs along with the levels of LL-37 and NETs products in the blood. Measurements will be repeat three months after the mainstay continuous positive airway pressure (CPAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old, with moderate to severe OSA (AHI ≥ 15/hour), and willing to participate in the study.

Exclusion Criteria:

* Under 20 years old, suffering from diseases or conditions that may affect immune function (e.g., tumors, chemotherapy, autoimmune diseases, diabetes, chronic kidney disease, etc.), or unwilling to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Moderate-to-Severe OSA
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
NET activity of neutrophils induced by PMA | From enrollment to receiving CPAP therapy for 3 months
  10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Neutrophils are isolated from peripheral blood and stimulated with PMA (phorbol 12-myristate 13-acetate) to induce the formation of NETs. The effects were tested with or without intermittent hypoxia (IH) treatment (1% O₂ for 35 minutes followed by 21% O₂ for 25 minutes per cycle, repeated for three cycles). The extent of NETs formation was assessed by confocal microscopy and images were exported as multi-channel TIFF files and analyzed using custom Python scripts (NumPy, scikit-image).
DNA-MPO (Myeloperoxidase) complex in plasma | From enrollment to receiving CPAP therapy for 3 months
  Description: 10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Plasma is collected and tested for DNA-MPO (Myeloperoxidase) complex by ELISA (Enzyme-linked immunosorbent assay).
LL-37 level in plasma | From enrollment to receiving CPAP therapy for 3 months
  10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Plasma is collected and tested for LL-37 by ELISA (Enzyme-linked immunosorbent assay).

OTHER OUTCOMES:
LL-37 in the supernatant of cultured neutrophils | From enrollment to receiving CPAP therapy for 3 months
  10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Neutrophils are isolated from peripheral blood and stimulated with PMA (phorbol 12-myristate 13-acetate) to induce the formation of NETs. Supernatant of cultured neutrophils are collected and tested for LL-37 by ELISA.
MPO (Myeloperoxidase) in the supernatant of cultured neutrophils | From enrollment to receiving CPAP therapy for 3 months
  10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Neutrophils are isolated from peripheral blood and stimulated with PMA (phorbol 12-myristate 13-acetate) to induce the formation of NETs. Supernatant of cultured neutrophils are collected and tested for MPO (Myeloperoxidase )by ELISA.
NE (Neutrophil elastase) in the supernatant of cultured neutrophils | From enrollment to receiving CPAP therapy for 3 months
  10 cc peripheral venous blood of participants will be collected at enrollment and 3 months after CPAP therapy (if received it). Neutrophils are isolated from peripheral blood and stimulated with PMA (phorbol 12-myristate 13-acetate) to induce the formation of NETs. Supernatant of cultured neutrophils are collected and tested for NE (Neutrophil elastase) by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol